CLINICAL TRIAL: NCT01169753
Title: Nuvigil in Treatment of Cancer-Related Fatigue in Chronic Myeloid Leukemia (CML) on Imatinib, Dasatinib, Nilotinib (or Any Other FDA Approved TKI for CML)
Brief Title: Nuvigil in Treatment of Cancer-Related Fatigue in Chronic Myeloid Leukemia Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow Enrollment
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Cephalon (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2009-0638; NCI-2011-00895 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-07-23; First posted 2010-07-26 (Estimated); Results first posted 2015-12-08 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-11

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Chronic Myeloid Leukemia; CML; Nuvigil; Armodafinil; Fatigue
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Fatigue | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Patients randomized to nonintervention will take a placebo every morning for 2 weeks.
  Interventions: Drug: Placebo
- Armodafinil (Experimental): Three 50 mg tablets orally every morning for 2 weeks.
  Interventions: Drug: Armodafinil

INTERVENTIONS:
Drug: Placebo — Oral tablet every morning for 2 weeks
  Arms: Placebo
Drug: Armodafinil — Three 50 mg tablets orally every morning for 2 weeks.
  Other Names: Nuvigil
  Arms: Armodafinil

SUMMARY:
The goal of this clinical research study is to learn if Nuvigil (armodafinil) can help to control fatigue in patients with CML. The safety of this drug will also be studied.

DETAILED DESCRIPTION:
The Study Drug:

Armodafinil is designed to help promote wakefulness in patients suffering from fatigue.

Study Groups:

If you are found to be eligible to take part in this study, you will take 3 tablets each day during Weeks 1, 2, 4, and 5. You will not take any tablets during Week 3.

You will be randomly assigned (as in the flip of a coin) to a study group. The tablets you receive will depend on which study group you are in. You will have an equal chance of being assigned to either group:

* If you are in Group 1, you will take armodafinil during Weeks 1 and 2 and a placebo during Weeks 4 and 5. A placebo is a tablet that looks like the study drug but has no active ingredients.
* If you are in Group 2, you will take a placebo during Weeks 1 and 2 and armodafinil during Weeks 4 and 5.

Neither you nor the study staff will know to which group you are assigned. However, if needed for your safety, the study staff will be able to find out what you are receiving at any time.

You will be given a fatigue diary and a drug diary. You will fill out the fatigue diary every day by answering 2 questions about fatigue. You will fill out the drug diary every day by writing when you take the study drug/placebo. You will return any unused drug/placebo at the end of Weeks 2 and 5.

At Week 5, you will be asked if you preferred the first period (Weeks 1 and 2 of the study) or the second period (Weeks 4 and 5 of the study). If your doctor thinks it is in your best interest and you are benefitting at this point, you will be able to continue taking the study drug and you will have additional study visits.

If you are one of the patients selected for the PK testing, the final results of the PK testing for your entire group will need to be completed before you can start the long term use of the study drug. If you take the study drug after Week 5, you will take 3 tablets every day for the rest of the time that you take the study drug.

Study Visits:

At the end of Weeks 1, 3, and 4:

* You will be asked about any symptoms that you may be having and about any other drugs that you may be taking.
* You will complete 2 questionnaires about fatigue and activity. It will take about 10 minutes to complete these questionnaires.
* Your blood pressure will be measured (Weeks 1 and 4 only).

At the end of Weeks 2 and 5:

* You will have a physical exam, including measurement of your weight and vital signs.
* You will complete the same questionnaires you completed at screening.
* Blood (about 1 teaspoon) will be drawn for routine tests.
* If you were selected for PK testing during screening, you will also have PK blood samples drawn at the end of Week 2 and Week 5.
* You will complete the series of tests that check your memory, motor skills, and thinking that you completed at screening.

At Weeks 10, 15, 20, and 25:

* You will be asked about any symptoms that you may be having and about any other drugs that you may be taking.
* You will complete the 2 questionnaires about fatigue and activity.
* Your blood pressure will be measured.

If you are not scheduled to come to MD Anderson at Weeks 1, 3, 4, 10, 15, 20, and 25, the procedures to be performed at these times can be performed at home. You will be called and asked the questions described in these visits. You will take 2 separate blood pressure measurements 5 minutes apart for each day and report results to the research staff over the telephone. If you choose to take your blood pressure measurements at home, you will be provided with a home blood pressure monitor at screening and taught how to use it. The monitor will be returned to study staff at the end of the study.

Length of Study:

You may continue taking the study drug as part of this study for up to 24 weeks. If you are benefiting after 24 weeks, you may continue taking the study drug off study. If you are one of the patients selected for the PK testing, the final results of the PK testing for your entire group will need to be completed before you can start the long term use of the study drug. You will be taken off study at any time if you have intolerable side effects or if the study doctor thinks it is in your best interest.

End of Treatment:

About 6 months after the end of Week 5, the following tests and procedures will be performed:

* You will complete the same questionnaires you completed at screening.
* You will complete the series of tests that check your memory, motor skills, and thinking that you completed at screening.
* Blood (about 1 teaspoon) will be drawn for routine tests.
* You will have a physical exam, including measurement of your weight and vital signs.

Follow-Up:

The study staff will call you about 30 days after your last dose of study drug and ask about any symptoms or complaints you may have had, as well as about any other drugs you may be taking. This call will last about 10 minutes.

This is an investigational study. Armodafinil is FDA approved and commercially available to help improve wakefulness in adults who experience excessive sleepiness. Its use in cancer-related fatigue is investigational.

Up to 60 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with CML on imatinib, dasatinib or nilotinib (or any other FDA approved tyrosine kinase inhibitor (TKI) for CML)
2. Must be >/= 18 years of age
3. Must have "fatigue worst" on The Brief Fatigue Inventory > or = 4
4. Women of childbearing potential (not surgically sterile or 2 years postmenopausal) must use a medically accepted method of contraception (refer to protocol for acceptable methods of contraception). Men not surgically sterile or who are capable of producing offspring must practice abstinence or use a barrier method of birth control. Both men and women must agree to continue use of this method for the duration of the study and for 30 days after participation in the study.
5. Informed consent must be signed
6. Patient should have at least a complete cytogenetic response (CCyR) sustained for the last 6 months
7. Patient should be receiving stable dose of TKI for at least 3 months (i.e. no increase or decrease in dose during this period) and should not have treatment interruptions for more than 7 consecutive days during this time period unless this was exclusively because of fatigue.
8. Females must have a negative serum pregnancy test within 48 hours prior to beginning treatment on this trial
9. Patient has an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2 at baseline

Exclusion Criteria:

1. History of hypersensitivity or allergy to armodafinil, modafinil or any component of the formulation of armodafinil.
2. History of or current seizures, glaucoma, major psychiatric diagnosis (psychiatric illness that required hospitalization), narcolepsy or Tourette's syndrome
3. History of severe headaches or increased agitation within the last 90 days prior to enrollment
4. History of clinically significant uncontrolled pulmonary or cardiac disease (uncontrolled is defined as patients requiring changes in dose and/or start of a new course of treatment in the last 30 days). This may include disease states as congestive heart failure, cardiac arrhythmias, coronary artery disease, chronic obstructive pulmonary disease and asthma)
5. Uncontrolled hypertension. Patients that have not been on a stable treatment dose for the past month or have a systolic blood pressure consistently (consistently is defined as 3 consecutive blood pressure readings within the last 30 days) greater than 150 mm Hg or diastolic pressure consistently greater than 85 mm Hg
6. History of fibromyalgia
7. History or current abuse of alcohol or drugs
8. Moderate to severe depression as measured on the Depression Anxiety Stress Scale (DASS-21)
9. If taking antidepressants, no changes in dose and/or no start of new course of treatment in the last 30 days
10. Currently taking psychostimulants (including appetite suppressants), L-Monoamine oxidases (MAO) inhibitors, anticoagulant therapy, anticonvulsant therapy or current consumption of alcohol within 8 hours of enrollment.
11. Current use of corticosteroids, stimulants, or other medications used to improve fatigue symptoms. Topical corticosteroids or occasional, intermittent doses of systemic steroids (e.g., for pre-medications, etc) are allowed
12. On clinical trials listing Armodafinil as a prohibited medication within the last 30 days of enrollment
13. Use of the following herbals or supplements for fatigue relief within the last 30 days (including dehydroepiandrosterone (DHEA), SAMe, ginkgo, ginseng, green, black or Chinese tea, ephedra (aka-ma-huang), popotillo and Mormon tea
14. Any coexisting medical condition or taking any concomitant medication that is likely to interfere with the safe administration of armodafinil
15. Hemoglobin < 8 gm/dl at time of enrollment
16. Albumin value 50% lower than the lower limit of normal
17. Evidence of hepatic impairment (total bilirubin > or = 2.5 times Upper limits of normal (ULN), serum glutamate pyruvate transaminase (SGPT) > or = 2.5 times ULN)
18. Evidence of renal impairment (serum creatinine > 2.5 times ULN)
19. If taking opioids, anxiolytics, and/or hypnotics, no changes in dose and/or no start of new course of treatment in the last 30 days
20. Patients who were ever in blast phase of CML
21. Female patients who are pregnant or breastfeeding
22. History of mitral valve prolapse documented by cardiac study.
23. Patients with history or current suicidal ideation
24. Currently taking strong cytochrome P450 3A4 (CYP3A4) inducers (including but not limited to phenobarbital, phenytoin, rifampin,and troglitazone); strong CYP3A4 inhibitors (including but not limited to ketoconazole, itraconazole, clarithromycin, ritonavir, indinavir, nelfinavir, saquinavir, nefazodone, telithromycin and grapefruit juice)
25. Patients who have been transplanted and are on immunosuppressive therapies that may interfere with TKI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-05; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Escalante, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: May 12, 2011 to December 4, 2012. All recruitment done at The University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: Study terminated early due to slow accrual.
Groups:
- Placebo: Oral placebo every morning for 2 weeks.
- Armodafinil: Armodafinil Three 50 mg tablets orally every morning for 2 weeks.
Period: Overall Study
Arm/Group | Placebo | Armodafinil
Started | 0 | 1
Completed | 0 | 0
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Armodafinil | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Number; unit: participants]
  <=18 years |  | 0 | 0
  Between 18 and 65 years |  | 1 | 1
  >=65 years |  | 0 | 0
Gender [Number; unit: participants]
  Female |  | 1 | 1
  Male |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With "Fatigue Worst" BFI Score
Description: Efficacy defined by "fatigue worst" score from the Brief Fatigue Inventory (BFI) after each 2-week treatment period, using a 0 - 10 scale with 10 being WORST level of fatigue.
Time Frame: After each 2 week treatment
Population: No analysis completed, study stopped due to slow accrual with only one participant.
Arm/Group | Placebo | Armodafinil
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event reporting collected through week 5 of period two which includes 2 two-week treatment periods and one week for washout phase.
Arm/Group | Placebo | Armodafinil
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=0) | Armodafinil (N=1)
Heart racing (Investigations) | 0 (0) | 1 (1)
Insomnia (General disorders) | 0 (0) | 1 (1)
Jittery feeling (General disorders) | 0 (0) | 1 (1)
Decreased appetite (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes